CLINICAL TRIAL: NCT01060553
Title: Pilot of Acupuncture to Improve Quality of Life in Veterans With TBI and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Samueli Institute for Information Biology (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPO 09-258
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-08

CONDITIONS: Post-traumatic Stress Disorders
Keywords: Post-traumatic stress disorders; Acupuncture; Quality of life; sleep disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): The treatment program consisted of 24 semi-individualized acupuncture treatments over 12 weeks. It combines front and back treatments to avoid point fatigue (tolerance due to frequent use). The front treat-ment uses 11 needles, bilateral at acupuncture points LR3, PC6, HT7, ST36, SP6, and one at Yintang; the back treatment uses 14 needles, bilateral at points GB20, and BL14, 15, 18, 20, 21, and 23. There are 15 other points from which the flexibly prescribed points could be chosen
  Interventions: Other: Acupuncture treatment
- wait list control (No Intervention): subjects were put on a wait list control. due to small numbers completing in both groups, the data from the wait list who completed acupuncture are combined with the experimental treatment group for analysis.

INTERVENTIONS:
Other: Acupuncture treatment — This project was initially designed as a randomized trial with one group receiving treatment and the other wait list control, with delayed treatment. Due to extremely high dropout and cancellations and failure to return for post assessment, a midpoint assessment was added. Analysis was done on pre and post measures of all subjects who completed at least the midpoint assessment. Due to the very small number of subjects in the wait list control, the ones who completed 6 or 12 weeks of acupuncture after the wait list were combined with the few who completed the initial acupuncture for a pre-post single group analysis. for those who completed both the 6 and 12 week measures, the latest one was selected for analysis
  Arms: Arm 1

SUMMARY:
The purpose of this study is to examine if acupuncture improves Post-Traumatic Stress Disorder symptoms among veterans who participated in Operations Enduring Freedom and Iraqi Freedom. This study will also examine the degree of veteran acceptance for acupuncture.

DETAILED DESCRIPTION:
Project Background: Acupuncture can be effective for many of the specific co-morbidities that make up war-related Trauma Spectrum Disorder in both TBI and PTSD patients, including pain, stress and anxiety, insomnia, somatic and post-operative pain. Recent studies find very large effect sizes (Cohen's D .85 to 1.4). Thus, there is good reason to believe that acupuncture will induce recovery across a number of trauma spectrum dysfunctions in patients with TBI and PTSD, at low cost and with little risk.

Project Objectives: The overall objective of this application is to determine the efficacy of adjunctive acupuncture for improving quality of life and function and alleviating co-morbidities associated with TBI and PTSD in service members injured in the current wars. The primary hypothesis of this study is: OIF/OEF veterans who screen positive for TBI or PTSD and are treated with a 12 week standard individualized acupuncture method will experience improved HRQL (as measured by the Veteran's SF-36) at 6, 12 and 24 week follow-up, compared to veterans randomly assigned to standard care alone.

Project Methods: This is a pilot study on veterans who screen positive for TBI or PTSD in the VA healthcare record, which is being submitted to obtain additional pilot data, confirmation of recruitment strategies, and information on non-participants . Frequency distribution and summary statistics for demographics and baseline variables will be presented by intervention group and for all subjects combined. Key demographic variables to be summarized are: age, gender, time to deployment, number of deployments, and diagnosis. Key baseline variables are: PTSD CAPS score, VSF-36, and ANAM score.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or positive screen test for PTSD.
* Combat veterans of Operation Iraqi Freedom or Operation Enduring Freedom conflicts.

Exclusion Criteria:

* Unable to travel to East Orange VA for 12 consecutive weeks, biweekly for treatment.
* Does not speak English.
* Acupuncture or CBT treatment within the previous six months.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Findley, MD PhD, Principal Investigator — East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ
Locations (1):
- East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 34 subjects were interviewed for consent. 15 were assigned to immediate treatment. 15 were assigned to wait list treatment. 2 did not meet inclusion criteria. 2 were assigned to case study.
Groups:
- Active Treatment: The treatment program consisted of 24 semi-individualized acupuncture treatments over 12 weeks. It combines front and back treatments to avoid point fatigue. The front treatment uses 11 needles, bilateral at acupuncture points LR3, PC6, HT7, ST36, SP6, and one at Yintang; the back treatment uses 14 needles, bilateral at points GB20, and BL14, 15, 18, 20, 21, and 23. There are 15 other points from which the flexibly prescribed points could be chosen
  Acupuncture treatment: Traditional Chinese theory explains acupuncture as a technique for balancing the flow of energy - believed to flow through pathways (meridians) in your body. Acupuncture involves the insertion of extremely thin, stainless steel, sterile needles in subcutaneous tissue or muscle at strategic points on your body which correspond to the acupuncture meridians. The Traditional Chinese Medicine (TCM) interview also includes looking at the tongue and feeling the pulse before deciding on all the points to be used.
- Wait List Control: this group was originall randomly assigned to a wait list control. due to severe recruitment and retention problems, data was collected in those willing to be treated after the wait list. this treatment data is combined with the original treatment group. this group received the same treatment, namely The treatment program consisted of 24 semi-individualized acupuncture treatments over 12 weeks. It combines front and back treatments to avoid point fatigue. The front treatment uses 11 needles, bilateral at acupuncture points LR3, PC6, HT7, ST36, SP6, and one at Yintang; the back treatment uses 14 needles, bilateral at points GB20, and BL14, 15, 18, 20, 21, and 23. There are 15 other points from which the flexibly prescribed points could be chosen
Period: Overall Study
Arm/Group | Active Treatment | Wait List Control
Started | 15 | 15
Completed | 6 (5 subjects completed more than half the sessions and midpoint outcome measures were obtained) | 5
Not Completed | 9 | 10
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: 24 semi-individualized acupuncture treatments over 12 weeks. The front treat-ment uses 11 needles, bilateral at acupuncture points LR3, PC6, HT7, ST36, SP6, and one at Yintang; the back treatment uses 14 needles, bilateral at points GB20, and BL14, 15, 18, 20, 21, and 23. There are 15 other points from which the flexibly prescribed points could be chosen
Arm/Group | Arm 1
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: SF-36
Description: global health functioning Mental component (MCS) and Physical component (PCS) subscales range from 0 to 100 with 100 being better; 50 is expected population average.
Time Frame: baseline, 6 or 12 weeks (latest available is used)
Population: due to very small numbers of completers in the acupuncture and the wait list control, the data from the wait list group who completed at least 6 weeks of treatment were combined with those initially assigned to treatment for a single group pre/post analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: The treatment program consisted of 24 semi-individualized acupuncture treatments over 12 weeks. It combines front and back treatments to avoid point fatigue (tolerance due to frequent use). The front treat-ment uses 11 needles, bilateral at acupuncture points LR3, PC6, HT7, ST36, SP6, and one at Yintang; the back treatment uses 14 needles, bilateral at points GB20, and BL14, 15, 18, 20, 21, and 23. There are 15 other points from which the flexibly prescribed points could be chosen
  Acupuncture treatment: This project was initially designed as a randomized trial with one group receiving treatment and the other wait list control, with delayed treatment. Due to extremely high dropout and cancellations and failure to return for post assessment, a midpoint assessment was added. Analysis was done on pre and post measures of all subjects who completed at least the midpoint assessment
Arm/Group | Arm 1
Number analyzed (Participants) | 11
units on a scale
  mcs pre treatment | 35.2 (10.7)
  mcs post treatment | 39.0 (12.6)
  pcs pre treatment | 41.2 (9.9)
  pcs post treatment | 44.5 (9.5)
Statistical Analysis 1: Comparison: Arm 1; for mcs; Test type: Superiority or Other; p = .15, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1; for pcs; Test type: Superiority or Other; p = .28, t-test, 2 sided

2. Secondary Outcome: Pittsburgh Sleep Index
Description: subscales range from 0 to 3 with higher being worse.
Time Frame: baseline, 6 or 12 weeks (latest available is used)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: The treatment program consisted of 24 semi-individualized acupuncture treatments over 12 weeks. It combines front and back treatments to avoid point fatigue. The front treatment uses 11 needles, bilateral at acupuncture points LR3, PC6, HT7, ST36, SP6, and one at Yintang; the back treatment uses 14 needles, bilateral at points GB20, and BL14, 15, 18, 20, 21, and 23. There are 15 other points from which the flexibly prescribed points could be chosen
  Acupuncture treatment: Traditional Chinese theory explains acupuncture as a technique for balancing the flow of energy - believed to flow through pathways (meridians) in your body. Acupuncture involves the insertion of extremely thin, stainless steel, sterile needles in subcutaneous tissue or muscle at strategic points on your body which correspond to the acupuncture meridians. The Traditional Chinese Medicine (TCM) interview also includes looking at the tongue and feeling the pulse before deciding on all the points to be used.
Arm/Group | Arm 1
Number analyzed (Participants) | 11
units on a scale
  sleep duration pre | 2.4 (0.7)
  sleep duration post | 2.1 (0.7)
  sleep disturbance pre | 2.4 (0.5)
  sleep distubance post | 1.7 (0.7)
  sleep latency pre | 2.6 (0.5)
  sleep latency post | 1.7 (1.2)
Statistical Analysis 1: Comparison: Arm 1; for sleep duration; Test type: Superiority or Other; p = .34, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1; for sleep disturbance; Test type: Superiority or Other; p = .001, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1; for sleep latency; Test type: Superiority or Other; p = .015, t-test, 2 sided

ADVERSE EVENTS:
Description: due to small numbers of completers in both groups, data from the wait list group who completed subsequent treatment were combined with those initially assigned to treatmen for a pre/post single group analysis
Groups:
- Arm 1: The treatment program will consist of 24 semi-individualized acupuncture treatments over 12 weeks. It combines front and back treatments to avoid point fatigue (tolerance due to frequent use). The front treat-ment uses 11 needles, bilateral at acupuncture points LR3, PC6, HT7, ST36, SP6, and one at Yintang; the back treatment uses 14 needles, bilateral at points GB20, and BL14, 15, 18, 20, 21, and 23. There are 15 other points from which the flexibly prescribed points could be chosen
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
very small numbers of subjects due to dropout and loss to followup. data from the wait list subjects who completed the intervention were combined with those initially assigned to treatment for a pre/post single group analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes